CLINICAL TRIAL: NCT00522639
Title: Determination of the Predictive Value of FDG-PET-CT Scans, Blood Proteins and Blood Cells for the Prognosis for Patients With Lung Cancer Receiving Concurrent Chemo-Radiation
Brief Title: Predictive Value of FDG-PET-CT Scans for Patients With Lung Cancer Receiving Concurrent Chemo-Radiation
Acronym: FDG-PET lung
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Dr. D.K.M. De Ruysscher, MAASTRO clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-02-117; TACIR
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Lung Cancer; SCLC; NSCLC
Keywords: lung cancer; FDG-PET-CT; blood proteins; prognose
MeSH Terms: conditions — Lung Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 18F-deoxyglucose (FDG) — contrast medium

SUMMARY:
The objective of the study is to investigate the evolution ofn 18F-deoxyglucose (FDG) uptake and the tumour characteristics determined in the plasma of patients with lung cancer of during and after concurrent radiotherapy and chemotherapy

DETAILED DESCRIPTION:
This translational research part is aiming to give more insights in the way radiation injury and tumour response develops.

It involves three parts:

1. Repetitive FDG-PET-CT scans in order to assess early tumour response monitoring.
2. Blood sampling before, during and after radiotherapy in order to find predictors for normal tissue injury and for tumour response.
3. Extra staining of tumour biopsies

The FDG-PET-CT scan with i.v. contrast gives information of the tumour metabolism and its morphology. Therefore, one extra FDG-PET-CT scans will be done during radiotherapy at day 8. Tumour response will be determined by FDG-PET-CT scans 3 months after radiotherapy.

Blood samples

1. Before radiotherapy, 12 millilitres of blood (EDTA tubes) will be taken according to serum protocol (appendix 5).
2. At day 7, day 14 during concurrent chemo-radiation, 7 days after the end of this treatment and 3 months and 9 months after the end of radiotherapy, 12 millilitres serum (EDTA tube) will be taken to investigate the evolution of the proteins [In the first place, plasma concentrations of osteopontin and soluble CA9 for hypoxia, CRP and IL-6 for inflammation, total and free VEGF for angiogenesis and total and cleaved cytokeratin 18 for necrosis/apoptosis will be determined] during and after treatment, for its kinetics may be important as predictive factors. Standard ELISA tests will be used to determine these levels.
3. Before radiotherapy, at day 7 and at day 14 during radiation, 7 days after the end of this treatment and 3 months and 9 months after the end of radiotherapy, 24 millilitres of blood (EDTA tubes) will be taken to investigate the evolution of circulating cells and their progenitors during and after treatment.

The tumour biopsies may be stained with markers for proliferation (e.g. KI 67), apoptosis (e.g. M30), hypoxia (e.g. CA 9, Glut 1 and 3) and others (e.g. EGFR and EGFRvIII), in order to correlate these measurements with response.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven non-small cell or small cell lung cancer UICC stage I-III (in case of small cell lung cancer: limited stage)
* WHO performance status 0-2
* Less than 10 % weight loss the last 6 months
* In case of previous chemotherapy, concurrent chemo-radiotherapy can start after a minimum of 21 days after the last chemotherapy course
* No recent (< 3 months) severe cardiac disease (arrhythmia, congestive heart failure, infarction)
* No active peptic oesophagitis
* Life expectancy more than 6 months
* Measurable cancer
* Willing and able to comply with the study prescriptions
* 18 years or older
* Not pregnant and willing to take adequate contraceptive measures during the study
* Have given written informed consent before patient registration
* No previous radiotherapy to the chest

Exclusion Criteria:

* Not non-small cell or small cell histology, e.g. mesothelioma, lymphoma
* Malignant pleural or pericardial effusion
* History of prior chest radiotherapy
* Recent (< 3 months) myocardial infarction
* Uncontrolled infectious disease
* Distant metastases (stage IV)
* Patients with active peptic oesophagitis in the last year
* Less than 18 years old
* Pregnant or not willing to take adequate contraceptive measures during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-10; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Tumour response, measured with FDG-PET-CT scans 3 months post-radiation. as a function of delta FDG uptake the first week during radiotherapy | 9 months post-radiation

SECONDARY OUTCOMES:
- Incidence of acute radiation-induced oesophagitis - Incidence of radiation-induced pulmonary toxicity 3 and 9 months post-radiation | 9 months post-radiation

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD PhD, Principal Investigator — MAASTRO, Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, MAASTRO, Maastricht, Limburg, Netherlands